CLINICAL TRIAL: NCT00742313
Title: Effect on Bleeding When Using FloSeal Matrix™ in Subjects Undergoing Endoscopic Vein Harvest (EVH)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No statistical differences on study endpoints between groups.
Sponsor: Duke University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00009897
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2013-11

CONDITIONS: Bleeding
Keywords: Endoscopic; saphenous; vein; harvest
MeSH Terms: conditions — Hemorrhage | interventions — FloSeal Matrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Arm A has FloSeal Matrix applied to EVH wound bed.
  Interventions: Biological: FloSeal Matrix
- Arm B (No Intervention): Arm B does not have FloSeal Matrix applied to EVH wound bed.

INTERVENTIONS:
Biological: FloSeal Matrix — 10 ml of FloSeal Matrix will be applied to the endoscopic wound bed.
  Other Names: FloSeal Hemostatic Matrix
  Arms: Arm A

SUMMARY:
This is a prospective, randomized trial to see in patients undergoing coronary artery bypass grafting and endoscopically-harvested greater saphenous vein, if using FloSeal Matrix in the endoscopically-harvested saphenous vein wound bed decreases bleeding and complications.

DETAILED DESCRIPTION:
Purpose of Study: The primary objective of this study is to determine if using a hemostatic agent (FloSeal Matrix™) in the tunnel of the endoscopically harvested Greater Saphenous vein will decrease bleeding from that site. Secondary objectives are to determine if there is a decrease in the infection-rate at the site of the vein-harvested leg where the FloSeal Matrix™ was used compared to the ones where FloSeal Matrix™ was not used.

Background and Significance: FloSeal Matrix™ is indicated in surgical procedures (other than ophthalmic) as an adjunct to hemostasis when control of bleeding by ligature or conventional procedures is ineffective or impractical. It works on wet, actively bleeding tissue and conforms to irregular wound surfaces. It is proven to control bleeding from oozing to pulsatile flow. The EVH wound bed is irregular and hemostasis is, at times, difficult to obtain using conventional procedures such as ligature or cautery.

Design and Procedures: This is a prospective, randomized clinical trial that compares the effects of applying FloSeal Matrix™ to the EVH wound bed to not applying FloSeal Matrix™ to the EVH wound bed.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a consent form that has been approved by the Institutional Review Board.
2. Be at least 18 years of age.
3. Scheduled to undergo coronary artery bypass grafting with EVH.
4. Be able to return to Duke University Medical Center for post-operative visit.

Exclusion Criteria:

1. Be participating concurrently in another clinical trial that involves an investigational drug or device that would interfere with this study.
2. Reported allergy to FloSeal Matrix™

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Lowe, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Duke Hospital identified as undergoing endovein harvest of their saphenous vein.
Pre-assignment Details: Once subjects were enrolled,randomization occurred on the day of surgery. Only subject who's surgery did not occur as scheduled may have been screen failed.
Groups:
- FloSeal Matrix: FloSeal Matrix applied to EVH wound bed.
- Non-FloSeal Matrix: FloSeal Matrix was not added to the wound bed
Period: Overall Study
Arm/Group | FloSeal Matrix | Non-FloSeal Matrix
Started | 25 | 19
Completed | 24 | 19
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- FloSeal: Arm A has FloSeal Matrix applied to EVH wound bed.
- Control: Arm B does not have FloSeal Matrix applied to EVH wound bed.
- Total: Total of all reporting groups
Arm/Group | FloSeal | Control | Total
Number analyzed (Participants) | 25 | 19 | 44
Age, Customized [Number; unit: Participants]
  Greater than 18 years | 25 | 19 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 24 | 15 | 39
Region of Enrollment [Number; unit: participants]
  United States | 25 | 19 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Decreased Bleeding
Description: The number of participants with less than expected bleeding (bleeding typically expected for the vein grafting procedure) at the surgical site. Blood was collected in the Blake drain of the EVH wound bed treated with FloSeal MatrixFloSeal Matrix™in the tunnel of the endoscopically harvested Greater Saphenous vein.
Time Frame: 14 days
Population: Six participants were not analyzed due to early termination of study
Measure: Number; unit: participants
Groups:
- FloSeal Matrix: Arm A has FloSeal Matrix applied to EVH wound bed.
Arm/Group | FloSeal Matrix | Control
Number analyzed (Participants) | 25 | 19
participants | 25 | 19

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/19
Other Adverse Events (participants affected / at risk) | 0/25 | 0/19

LIMITATIONS AND CAVEATS:
This study was terminated early

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No